CLINICAL TRIAL: NCT06964802
Title: The Effect of Cold Salt Water Foot Bath on the Development Of Chemotherapy-Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tuba Eryiğit (Other)
Responsible Party: Sponsor-Investigator, Tuba Eryiğit, Research assistant/Specialist nurse, Istanbul Topkapi University
Organization: Istanbul Topkapi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulTopkapiU
Record Dates: First submitted 2025-04-24; First posted 2025-05-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Patients; Chemotherapy Induced Peripheral Neuropathy (CIPN); Paclitaxel-induced Peripheral Neuropathy
Keywords: Chemotherapy-Induced Peripheral Neuropathy; Cold Salt Water; Foot Bath; Breast Cancer; Paclitaxel
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Cold salt water foot bath group) (Experimental): During the three hours of paclitaxel treatment, 30 minutes of salt cold water foot bath application four times as 10 minutes break Patients will be evaluated with Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) and Chemotherapy Induced Peripheral Neuropathy Assessment Tool (CIPNAT) before the following chemotherapy cycle after the application of salt cold water foot bath during each cycle. These evaluations will be completed after 12 cycles and patients will be evaluated with CTCAE v5.0 and CIPNAT for a total of 12 times. In addition, all patients will be evaluated with vibration and monofilament test at the end of the 12th cycle.
  Interventions: Other: Cold salt water foot bath
- Group B (Cold unsalted water foot bath group) (Active Comparator): During the three hours of paclitaxel treatment, 30 minutes unsalted cold water foot bath application four times as 10 minutes break Patients will be evaluated with Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) and Chemotherapy Induced Peripheral Neuropathy Assessment Tool (CIPNAT) before the following chemotherapy cycle after the application of unsalted cold water foot bath during each cycle. These evaluations will be completed after 12 cycles and patients will be evaluated with CTCAE v5.0 and CIPNAT for a total of 12 times. In addition, all patients will be evaluated with vibration and monofilament test at the end of the 12th cycle.
  Interventions: Other: Cold water foot bath
- Group C (control group) (No Intervention): Patients in this group will be given general information about the care guidelines for chemotherapy patients at the clinic where they receive treatment. This information will be provided once. At the end of the study, patients in the control group will be offered a choice of two application methods, and the method they choose will be applied to them in the same way as to Groups A and B.
  Group C patients will be evaluated with Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) and Chemotherapy Induced Peripheral Neuropathy Assessment Tool (CIPNAT) before each chemotherapy cycle at the same time with Group A and B patients. In addition, all patients will be evaluated with vibration and monofilament test at the end of the 12th cycle.

INTERVENTIONS:
Other: Cold salt water foot bath — The application of 175 grams of salt to cold water at a constant 22 degrees
  Arms: Group A (Cold salt water foot bath group)
Other: Cold water foot bath — Constant 22 degree cold water application
  Arms: Group B (Cold unsalted water foot bath group)

SUMMARY:
This prospective, randomised, controlled study was designed to evaluate the effectiveness of salt and unsalted cold water foot baths in preventing chemotherapy-induced peripheral neuropathy (CIPN) in patients receiving paclitaxel. The study's sub-objectives were to minimise the development of CIPN, reduce its severity and incidence of symptoms, and minimise its impact on daily life and activities.

Hypothesis(es):

H1: Salt cold water foot bath affects the development of chemotherapy-induced peripheral neuropathy.

H2: There is an effect of unsalted cold water foot bath on the development of chemotherapy-induced peripheral neuropathy.

H3: The effects of salt and unsalted cold water foot baths on the development of chemotherapy-induced peripheral neuropathy.

H4: Salt and unsalted cold water foot baths are more effective than standard clinical care in the development of chemotherapy-induced peripheral neuropathy.

Researchers will compare the salt cold water with the unsalted cold water, unsalted cold water and control group to determine whether the salt cold water has an effect on CIPN.

The experimental group and active comparator participants will continue the application for 12 cycles (12 weeks) of paclitaxel. The application will be applied by researcher Tuba Eryiğit. In addition, before each application for 12 weeks, the severity of CIPN, its effect on daily life and grade will be evaluated.

The control group will continue clinical routine care applications for 12 cycles (12 weeks). In addition, the severity of CIPN, its effect on daily life and grade will be evaluated before each treatment in the same way as the experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over.
* Conscious
* Speaking and understanding Turkish
* The diagnosis was breast cancer
* Those who will receive paclitaxel chemotherapy
* These are patients who answered 'no' to the 'A' section of the CIPNAT scale

Exclusion Criteria:

* Responding to the vibration test (if the practitioner does not feel the vibration when the patient says they feel the vibration, it means that neuropathy is present)
* Feeling pressure in one or none of the three areas on the plantar surface of the foot according to the monofilament test
* Previous chemotherapy-associated peripheral neuropathy
* Diagnosed with diabetes
* Open wounds or skin ulcers on the foot
* With peripheral and central nervous system disease
* Peripheral vascular disease,
* Patients with bone or soft tissue metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
To prevent the development of chemotherapy-associated peripheral neuropathy in patients | This was at the end of the 12th week of paclitaxel treatment.
  Patients who respond 'No' to part A of the CIPNAT scale and who do not respond to the monofilament and vibration tests will be considered free of chemotherapy-related peripheral neuropathy.

SECONDARY OUTCOMES:
If you are experiencing chemotherapy-related peripheral neuropathy, the symptoms should be mild, occur less frequently and have a minimal impact on your daily life and activities. | This was at the end of the 12th week of paclitaxel treatment.
  A score close to 0 on the Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) scale, which ranges from 0 to 140, and a grade close to 1 on the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 scale, which grades from 1 to 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpaşa Numune Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All participant responses and personal information will be used for scientific purposes only.